CLINICAL TRIAL: NCT04158375
Title: Molecular Mechanisms of Exercise Benefits to Insulin Resistant People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Consultant, Division of Endocrinology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-006273; 1R01AG062859-01A1 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Insulin Resistance; Obesity
Keywords: Resistance Exercise
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Insulin Resistant Exercise Group (Experimental): Resistance (RE) training will be performed 4 days per week using a combination of upper and lower body exercises at 8-12 repetitions per set. Resistance training will be performed using a combination of upper and lower body exercises using machine and free weights. Upper body exercises are chest press, incline press, seated row, lat pull down, triceps extension, biceps curl and lateral raises. Major muscle groups for upper body exercises will include chest (pectoralis major and minor), arm (biceps and triceps), shoulder (deltoids) and back (latissimus dorsi and rhomboids). Lower body exercises are leg press, lunge (with body weight progressing to dumbbells), seated leg extension, seated leg curl, calf raises and abdominal crunches. Major muscle groups for the lower body exercises will be thighs (quadriceps and hamstrings), calves (gastrocnemius and soleus) and core (rectus abdominus and obliques).
  Interventions: Behavioral: Resistance Exercise
- Insulin Resistant Control Group (No Intervention): Participants in this group will perform no exercise for the 3 month study period.
- Insulin Sensitive Lean Group (No Intervention): Participants in this group will have a baseline study for comparison to the insulin resistant groups.

INTERVENTIONS:
Behavioral: Resistance Exercise — Resistance (RE) training will be performed 4 days per week using a combination of upper and lower body exercises at 8-12 repetitions per set. Participants will complete 2 progressing to 4 sets of 8 to 12 repetitions per exercise, with 1 minute rest between sets. Participants will warmup for 5 minutes on a treadmill, cycle ergometer or elliptical at ~50% VO2 peak then begin resistance training. Resistance will be performed 4 days per week with lower body exercise on Monday and Thursday, and upper body on Tuesday and Friday. Wednesdays are a rest day. Participants will begin at 2 sets per exercise on weeks 1 and 2, then 3 sets for week 3, and 4 sets for weeks 4 to 12.
  Arms: Insulin Resistant Exercise Group

SUMMARY:
This proposal will investigate the underlying mechanisms of enhanced insulin sensitivity and improvement of muscle loss and performance in insulin resistant people by resistance exercise training. Based on the investigator's preliminary data, they hypothesize that the key regulators of health benefits of resistance training are two genes: PGC-1a4 and PPARB;, and that the increased expression of these genes following resistance training facilitates storage of glucose in muscle and enhances its utilization for the energy need of muscle for contraction as well as enhancing muscle mass and performance. The investigators will also determine whether resistance training can reduce the higher oxidative stress in insulin resistant humans and improve their muscle protein quality.

DETAILED DESCRIPTION:
Identification of the molecular regulatory points of exercise benefits is of high national priority because of the opportunity to develop targeted novel therapeutics benefiting populations suffering from inactivity-related health problems, including T2DM and pre-diabetes, characterized by insulin resistance (IR). IR is most prevalent in the older population associated with sarcopenia. The investigators propose a novel metabolic regulatory role of PGC-1α4 (α4), a hypertrophy gene, enhanced by resistance exercise (RE). Based on substantial preliminary data, the investigators hypothesize that α4, in cooperation with PPARβ (Rβ), promotes muscle glycolysis and insulin sensitivity (IS) as well as increasing muscle mass and performance. Based on their novel preliminary data, they will also investigate whether by deacetylation of glycolytic proteins, RE enhances muscle glycolytic capacity. Rβ also reduces oxidative stress that not only enhances IS but also contributes to other health benefits. New mRNA based data indicates that RE reduces protein degradation which will be investigated in the current proposal. The investigators will determine whether 3 months of RE training enhances insulin sensitivity and muscle performance and mass in IR people through pathways of enhanced glycolysis, deacetylation of glycolytic proteins reducing protein degradation and enhancing synthesis and ameliorating oxidative stress. They will study 48 IR people 50-75 yrs before and after 3 months of either 4-times/week resistance training or sedentary life and compare them with lean IS people. They will collect vastus lateralis muscle biopsy samples before and after an acute exercise bout and following a mixed meal to measure markers of glycolysis, energy metabolites, glycogen synthase, glycogen content, α4, Rβ, insulin signaling proteins and proteome analysis. They will also measure markers of oxidative stress including 8-OXO-dg (measure of DNA damage), oxidative damage to proteins and subsequent muscle protein degradation, which they hypothesize is reduced by increased anti-oxidant effect of Rβ with RE training. They also will use in vivo labeling of specific muscle proteins utilizing stable isotope labeled tracers to determine whether α4 induced muscle hypertrophy occurs not only by reducing degradation but also by enhancing contractile protein synthesis. These studies will render the necessary mechanistic explanation on how RE enhances IS, glycolysis, reduces oxidative stress and promote muscle performance and mass in IR people, thus substantially contributing to health and life span.

ELIGIBILITY:
Inclusion criteria

* age 50-75yrs
* BMI 30-38kg/m2
* hip to waist ratio of >0.85 in women and 1.0 in men
* fasting glucose ≥100-140mg/dl

Lean Group

* age 50-75 years
* hip to waist ratio of <0.76 in women and 0.90 in men
* fasting glucose of <100mg/dl.

Exclusion criteria for the study are as follows:

* Coronary artery disease or heart failure.
* Participation in a structured exercise program >2 days per week
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  * Inpatient psychiatric treatment in the past 6 months
  * Presence of a known adrenal disorder
  * Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
  * Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
  * Active gastroparesis
  * If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
  * Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L); testing required within three months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
  * Abuse of alcohol or recreational drugs
  * Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis).
  * Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg) at the time of screening.
  * Oral steroids
  * A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
  * Restrictions on Use of Other Drugs or Treatments:
  * Medications that may impact study end points such as mitochondrial biology eg. beta blockers
  * Anti-hyperglycemic drugs including metformin
  * Any other medication that the investigator believes is a contraindication to the subject's participation.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Sreekumaran Nair, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pataky MW, Heppelmann CJ, Sevits KJ, Asokan AK, Kumar AP, Klaus KA, Dasari S, Kunz HE, Strub MD, Robinson MM, Coon JJ, Lanza IR, Adams CM, Nair KS. Aerobic and resistance exercise-regulated phosphoproteome and acetylproteome modifications in human skeletal muscle. Nat Commun. 2025 Jul 1;16(1):5700. doi: 10.1038/s41467-025-60049-0. PMID 40595512
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Resistant Exercise Group: Resistance (RE) training will be performed 4 days per week using a combination of upper and lower body exercises at 8-12 repetitions per set. Resistance training will be performed using a combination of upper and lower body exercises using machine and free weights. Upper body exercises are chest press, incline press, seated row, lat pull down, triceps extension, biceps curl and lateral raises. Major muscle groups for upper body exercises will include chest (pectoralis major and minor), arm (biceps and triceps), shoulder (deltoids) and back (latissimus dorsi and rhomboids). Lower body exercises are leg press, lunge (with body weight progressing to dumbbells), seated leg extension, seated leg curl, calf raises and abdominal crunches. Major muscle groups for the lower body exercises will be thighs (quadriceps and hamstrings), calves (gastrocnemius and soleus) and core (rectus abdominus and obliques). Participants will complete 2 progressing to 4 sets, with 1 minute rest between sets. Participants will warmup. Resistance will be performed 4 days per week with lower body exercise on Monday and Thursday, and upper body on Tuesday and Friday. Wednesdays are a rest day. Participants will begin at 2 sets per exercise on weeks 1 and 2, then 3 sets for week 3, and 4 sets for weeks 4 to 12.
Period: Overall Study
Arm/Group | Insulin Resistant Exercise Group | Insulin Resistant Control Group | Insulin Sensitive Lean Group
Started | 33 | 16 | 9
Completed | 33 | 13 | 9
Not Completed | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Resistant Exercise Group | Insulin Resistant Control Group | Insulin Sensitive Lean Group | Total
Number analyzed (Participants) | 33 | 13 | 9 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 10 | 4 | 37
  >=65 years | 10 | 3 | 5 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 7 | 5 | 29
  Male | 16 | 6 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 32 | 12 | 8 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 33 | 13 | 9 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 33 | 13 | 9 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Strength
Description: Change in 1RM normalized to lean mass
Time Frame: Baseline and 3 Months
Population: Only longitudinal arms were analyzed since this is a measure of change between baseline and 3 months (Insulin Resistant Exercise Group vs Insulin Resistant Control Group). The Insulin Sensitive Lean Group was only for baseline comparisons.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Insulin Resistant Exercise Group: Resistance (RE) training will be performed 4 days per week using a combination of upper and lower body exercises at 8-12 repetitions per set. Resistance training will be performed using a combination of upper and lower body exercises using machine and free weights. Upper body exercises are chest press, incline press, seated row, lat pull down, triceps extension, biceps curl and lateral raises. Major muscle groups for upper body exercises will include chest (pectoralis major and minor), arm (biceps and triceps), shoulder (deltoids) and back (latissimus dorsi and rhomboids). Lower body exercises are leg press, lunge (with body weight progressing to dumbbells), seated leg extension, seated leg curl, calf raises and abdominal crunches. Major muscle groups for the lower body exercises will be thighs (quadriceps and hamstrings), calves (gastrocnemius and soleus) and core (rectus abdominus and obliques).
  Resistance Exercise: Resistance (RE) training will be performed 4 days per week using a combination of upper and lower body exercises at 8-12 repetitions per set. Participants will complete 2 progressing to 4 sets of 8 to 12 repetitions per exercise, with 1 minute rest between sets. Participants will warmup for 5 minutes on a treadmill, cycle ergometer or elliptical at ~50% VO2 peak then begin resistance training. Participants will begin at 2 sets per exercise on weeks 1 and 2, then 3 sets for week 3, and 4 sets for weeks 4 to 12.
Arm/Group | Insulin Resistant Exercise Group | Insulin Resistant Control Group
Number analyzed (Participants) | 32 | 15
Ratio | 0.37 (0.31) | -0.2 (0.32)

2. Primary Outcome: Change in Insulin Sensitivity
Description: Difference from baseline and 3 months of the insulin area on under the curve - A measure of insulin sensitivity as measured during an oral meal tolerance test - Time points (-20, 0, 10, 20, 30, 60, 90, 150, 240 minutes)
Time Frame: Baseline and 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μIU*min/mL
Arm/Group | Insulin Resistant Exercise Group | Insulin Resistant Control Group
Number analyzed (Participants) | 32 | 15
μIU*min/mL | -743.7 (2292) | -105.7 (2015)

3. Primary Outcome: Change in Lean Mass
Description: Change in body lean mass as measured by DEXA scan
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Insulin Resistant Exercise Group | Insulin Resistant Control Group
Number analyzed (Participants) | 32 | 15
grams | 542 (1526) | -377 (1348)

4. Secondary Outcome: Change in Fat Percentage
Description: Change in body fat percentage as measured by DEXA scan
Time Frame: Baseline and 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Insulin Resistant Exercise Group | Insulin Resistant Control Group
Number analyzed (Participants) | 32 | 15
Percentage | -0.89 (1.01) | 0.12 (1.14)

ADVERSE EVENTS:
Time Frame: Baseline to the end of intervention (3 months)
Description: Only longitudinal arms were monitored/assessed for adverse events (Insulin Resistant Exercise Group vs Insulin Resistant Control Group). The Insulin Sensitive Lean Group was only for baseline comparisons; there was no follow up and no intervention therefore adverse events were not monitored/assessed in the Insulin Sensitive Lean Group.
Arm/Group | Insulin Resistant Exercise Group | Insulin Resistant Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/15
Other Adverse Events (participants affected / at risk) | 0/32 | 0/15

LIMITATIONS AND CAVEATS:
There are no limitations or caveats at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT04158375/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04158375/ICF_001.pdf